CLINICAL TRIAL: NCT04395768
Title: Therapies to Prevent Progression of COVID-19, Including Hydroxychloroquine, Azithromycin, Zinc, Vitamin D, Vitamin B12 With or Without Vitamin C, a Multi-centre, International, Randomized Trial: The International ALLIANCE Study
Brief Title: International ALLIANCE Study of Therapies to Prevent Progression of COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Integrative Medicine, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Alliance-COVID19
Record Dates: First submitted 2020-05-18; First posted 2020-05-20 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: COVID19
Keywords: COVID19; hydroxychloroquine; azithromycin; zinc; Vit-D3; B12; C
MeSH Terms: conditions — COVID-19 | interventions — Ascorbic Acid; Hydroxychloroquine; Azithromycin; Cholecalciferol; Vitamin B 12

STUDY DESIGN:
Intervention Model Description: randomized investigator-blinded controlled
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants not blinded as they will know whether they are receiving the comparator vitamin c (either IVC) or oral in addition to treatments in the control group; outcomes assessor / investigators conducting statistical analysis will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin C (Experimental): Participants will receive vitamin C in addition to active comparator treatment:
  Inpatients: IV Vitamin C (Sodium Ascorbate) 50mg/kg every 6hrs on day 1 followed by 100mg/kg every 6hrs (4x per day; 400mg/kg/day) for 7 days (average 28g/day; maximum dose of 50g/24hrs for those weighing more than 125kg). Can be converted to 1 gram three times per day PO on hospital discharge) Outpatients: Vitamin C Outpatient trial: 200mg/kg x1 IV, then 1 gram PO three times per day for 7 days;
  Plus Active Comparator treatment:
  Hydroxychloroquine Hydroxychloroquine 400mg (2x200mg) PO for 1 day, followed by 200mg PO per day for 6 days Azithromycin 500 mg PO on day 1 followed by 250 mg PO once daily for 4 days Zinc Citrate 30mg elemental zinc PO daily Vitamin D3 5,000iu PO daily for 14 days Vitamin B12 (Methylcobalamin) 500mcg PO daily for 14 days
  Interventions: Dietary Supplement: Vitamin C; Drug: Hydroxychloroquine; Drug: Azithromycin; Dietary Supplement: Zinc Citrate; Dietary Supplement: Vitamin D3; Dietary Supplement: Vitamin B12
- Control (Active Comparator): Hydroxychloroquine Hydroxychloroquine 400mg (2x200mg) PO for 1 day, followed by 200mg PO per day for 6 days Azithromycin 500 mg PO on day 1 followed by 250 mg PO once daily for 4 days Zinc Citrate 30mg elemental zinc PO daily Vitamin D3 5,000iu PO daily for 14 days Vitamin B12 (Methylcobalamin) 500mcg PO daily for 14 days
  Interventions: Drug: Hydroxychloroquine; Drug: Azithromycin; Dietary Supplement: Zinc Citrate; Dietary Supplement: Vitamin D3; Dietary Supplement: Vitamin B12

INTERVENTIONS:
Dietary Supplement: Vitamin C — In addition to the active comparator, which is a combination of 2 drugs and 3 dietary supplements, the experimental treatment arm will also receive Vitamin C (intravenous or oral)
  Other Names: Sodium ascorbate
  Arms: Vitamin C
Drug: Hydroxychloroquine — Active comparator group will receive: a combination of 2 drugs and 3 dietary supplements
  Other Names: Plaquenil
Drug: Azithromycin — Active comparator group will receive: a combination of 2 drugs and 3 dietary supplements
  Other Names: Z-Pak; Zithromax
Dietary Supplement: Zinc Citrate — Active comparator group will receive: a combination of 2 drugs and 3 dietary supplements
Dietary Supplement: Vitamin D3 — Active comparator group will receive: a combination of 2 drugs and 3 dietary supplements
  Other Names: Cholecalciferol
Dietary Supplement: Vitamin B12 — Active comparator group will receive: a combination of 2 drugs and 3 dietary supplements
  Other Names: Methylcobalmin

SUMMARY:
COVID-19 is a global pandemic. So far encouraging results have been shown in different parts of the world with the utilisation of hydroxycloroquine, zinc, and azithromycin, and early studies into some of these, plus some with Vitamin C, have also proven beneficial. Vitamin D levels have also been shown to be an important indicator to the severity of symptoms in COVID-19 patients.

DETAILED DESCRIPTION:
Study Design

Type of study A multi-centre, open-label, randomized controlled trial evaluating the efficacy and safety of therapy with azithromycin, hydroxychloroquine, zinc, vitamin D3/B12 and IV vitamin C compared with azithromycin, hydroxychloroquine, zinc, vitamin D3/B12 in participants with COVID-19.

Expected number of participants The sample size for the study is a minimum of 100 participants in each arm. However, this sample size may change as this trial has an adaptive design.

Allocation procedure Randomization: Eligible patients that have provided informed written consent will be randomized by independent researcher. Randomization will be in randomly permuted blocks (undisclosed sizes to maintain concealment of allocation). The allocation will be communicated to site personnel and participants will be made aware of their assignment. It is not practical to use placebo in this trial.

Stratification: randomization will be stratified by site and age (65 years or younger, over 65 years of age).

Duration of the study period for each subject Participants will be followed for 45 days from the time of randomization. Data of events occurring during hospital will be obtained from hospital records supplemented by a telephone call or follow up at 7-10 days and at 45 days after randomization.

Adaptive design features

Adaptive intervention arms: The Steering Committee will keep abreast of other ongoing trials and if other promising interventions emerge, may recommend adding (or replacing) one arm with the new promising intervention.

Adaptive sample size: Sample size calculations are based on disease progression rates that are not well known. The investigators remain flexible, and the Data Safety Committee (DSMC) will be monitoring the possibility that the assumptions for sample size calculations may be modified with emerging information from this trial or other ongoing trials. If recruitment is going well, the steering committee may decide to extend recruitment as long as the independent DSMC does not terminate the trial for clear evidence of efficacy, futility (low probability) to detect a clinically meaningful difference (e.g. a 20% RRR in events) or concerns about safety.

Study Procedures Direct electronic data entry will be utilized in this trial. The investigators will use Redcap platform and software (www.project-redcap.org).

Consenting process Due to the stringent measures in infection control in hospitals, digitalised consent will be obtained instead of written consent on paper. Be this preferably from the patient or his legal representative. All patients will be in strict contact and droplet precautions and there may be an imperative to minimise use of personal protective equipment (PPE) by staff due to resource limitations.

The consenting process will be as follows:

* The clinical team will inform a potential participant in the trial that an investigator will contact them
* To minimise PPE use, the investigator will make telephone contact with the patient. If an interpreter is required for the consent discussion, this will be by the telephone interpreter service. An informed consent discussion will be held with each participant by a site investigator or their delegate.
* The Patient Information Sheet and Consent form (PICF) will be emailed to the patient or the clinical team will take it into the room for viewing by the patient. These documents will be left in the patient's room
* The participant will be given time to ask questions and consider whether to participate in the research.
* Verbal consent will be recorded in both the participant's medical record and study consent form. This will state that the terms and conditions were all read and agreed to and all questions asked were answered. The full PICF, including the signed consent page (by the investigator), will be uploaded into the electronic database.
* If the patient is too unwell or is unable to use a digital device, to personally give consent, written consent can be obtained from their next of kin, or other adult family members, or partner or legal representative.
* The following day, the investigator or clinical team will verbally confirm with the participant that they have consented to participate. A copy of the signed consent form will then either be emailed to the participant or sent via post. The participant, their next of kin or legal representative will send a return email confirming their consent.

Interventions

Blinding: Participants and healthcare providers will not be blinded to treatment. To account for this, the investigators have objective outcome definitions to minimize the opportunity for bias to influence event assessment.

Consenting participants will be randomized to receive therapy with azithromycin, hydroxychloroquine, zinc, Vitamin D3/B12 and IV vitamin C or azithromycin, zinc and hydroxychloroquine, Vitamin D3/B12.

For further details see: Arms & Interventions

The investigators will place no constraints for treating physicians on the therapies with respect to usual care. The investigators will document information on all key co-interventions, including information on drugs at the time of randomization and post randomization /during hospitalization.

Data collection The investigators will collect participant sex, age, disease severity, comorbidities (smoking, diabetes, heart disease, lung disease, immunosuppression, etc.), other medications, and trial outcomes.

Participants in this trial will be swabbed (nasal and/or oral) on approximately days 0, 3 and 7 for quantitative polymerase chain reaction (PCR) assessment of viral titre.

Study Outcomes For details see primary & secondary outcome section.

In addition, the investigators will collect data on:

WHO Master Protocol ordinal score at day 15:

1. Not hospitalized, no limitations on activities
2. Not hospitalized, limitation on activities;
3. Hospitalized, not requiring supplemental oxygen;
4. Hospitalized, requiring supplemental oxygen;
5. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
6. Hospitalized, on invasive mechanical ventilation or ECMO;
7. Death.

Secondary safety outcomes

* QTc prolongation (>500ms) 24 hours following initial dose of study drugs
* Serious ventricular arrhythmia (including ventricular fibrillation) or sudden unexpected death in hospital
* Any of the following adverse events in first 10 days from enrolment.
* Diarrhoea - grade 2 or greater
* Nausea - grade 2 or greater
* Vomiting - grade 2 or greater

Statistical Considerations

Sample size calculation The minimum sample size required is N=100 in each intervention arm in order to have 80% statistical power to detect a 30% relative risk reduction (RRR) in the proportion progressing to mechanical ventilation or death, assuming a standard-of-care risk of progression of 30%. Since participants will be hospitalized, a minimal (<1%) loss to follow-up is assumed.

Statistical analysis methods The primary analysis of efficacy will be conducted under the intention-to-treat principle; all randomized participants will be included in the analyses. All results will be analyzed with 2-sided level of significance of 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Provision of informed consent in writing, can be electronic
3. Diagnosis of active COVID-19

Exclusion Criteria:

1. Known G6PD deficiency
2. Contra-indication to hydroxychloroquine, azithromycin or Vitamin C: allergy to study interventions, epilepsy, serious hearing or visual problems, history of severe depression, calcium oxalate stones, advanced liver disease, pregnancy or lactating
3. Already receiving chloroquine, azithromycin, >3 grams Vitamin C daily or an experimental antiviral
4. History of fever (e.g. night sweats, chills) and/or acute respiratory infection (e.g. cough, shortness of breath, sore throat) of more than 7 days' duration. Note, if study numbers not quickly reached, the investigators may decide to include those with symptoms of longer than 7 days
5. Calculated creatinine clearance of < 30 mL/minute
6. Baseline ECG showing: QTc ≥470 for males, QTc ≥480 for females
7. Receipt of a drug known to increase QTc: quetiapine, amiodarone, sotalol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Symptoms | once daily for 15 days since enrollment/baseline at admission to hospital
  Composite measure: Change in severity and duration of symptoms
Length of hospital stay | at 15 and 45 days since admission/ enrolment
  total number of days in hospital since admission
invasive mechanical ventilation or mortality | any time within 15 days from enrolment
  need for invasive mechanical ventilation or mortality within 15 days from enrolment

SECONDARY OUTCOMES:
Mortality | 15 and 45 days since enrolment
  Death
mechanical ventilation | at 15 and 45 days since enrolment
  need for and number of days of invasive mechanical ventilation, in case of no need for mechanical ventilation: days=0
oxygen | 15 and 45 days since enrolment
  need for and number of days for humidified high-flow oxygen
ICU | 15 and 45 days since enrolment
  admission to ICU (intensive care unit)
days in hospital | 15 and 45 days since enrolment
  days in hospital
days in ICU | 15 and 45 days since enrolment
  days in ICU
renal replacement therapy | 15 and 45 days since enrolment
  need for and days of renal replacement therapy
Extracorporeal support | 15 and 45 days since enrolment
  need for and days of Extracorporeal support

CONTACTS AND LOCATIONS:
Overall Officials: Karin Ried, PhD, Principal Investigator — National Institute of Integrative Medicine, Australia
Locations (1):
- National Institute of Integrative Medicine, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No